CLINICAL TRIAL: NCT05880758
Title: Impact of Yo-Yo Sleep on Cardiometabolic Health
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Icahn School of Medicine at Mount Sinai (Other); University of Colorado, Denver (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Marie-Pierre St-Onge, Associate Professor, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: AAAU3694; R35HL155670 (NIH)
Record Dates: First submitted 2023-05-17; First posted 2023-05-30 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Cardiometabolic Syndrome; Obesity
Keywords: Sleep; Circadian Rhythms; Cardiometabolic Health
MeSH Terms: conditions — Metabolic Syndrome; Obesity

STUDY DESIGN:
Intervention Model Description: 3-arm, parallel study design
Who Masked: Outcomes Assessor
Masking Description: Statistician will be blinded to intervention allocation; blinding of study participants is not possible due to the intervention type.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Stable Adequate Sleep (SAS) (Active Comparator): Participants will go to bed and wake up at the same time every night, maintaining adequate sleep duration.
  Interventions: Behavioral: Sustained Adequate Sleep (SAS)
- ISS_Alone (Experimental): Intermittent short sleep (ISS) 5 nights of 5.5 hours time in bed 2 nights of 9.5 hours time in bed with advanced bedtimes and delayed wake times
  Interventions: Behavioral: Intermittent Short Sleep (ISS)
- ISS_SJL (Experimental): Intermittent short sleep with short jetlag (SJL) 5 nights of 5.5 hours time in bed 2 nights of 9.5 hours time in bed with constant bedtimes and delayed wake times
  Interventions: Behavioral: Intermittent Short Sleep (ISS); Behavioral: Social Jetlag (SJL)

INTERVENTIONS:
Behavioral: Intermittent Short Sleep (ISS) — Restricted sleep duration of <5.5 h/night for 5 nights (SR) followed by 2 nights of 9.5 hours of time in bed (TIB) (recover sleep) each week.
  Other Names: ISS
  Arms: ISS_Alone; ISS_SJL
Behavioral: Social Jetlag (SJL) — 2-hour delayed sleep timing.
  Other Names: SJL
  Arms: ISS_SJL
Behavioral: Sustained Adequate Sleep (SAS) — Goal of ≥7 hours of sleep/night with 8 hours of time in bed (TIB).
  Other Names: SAS
  Arms: Stable Adequate Sleep (SAS)

SUMMARY:
The goal of this clinical trial is to test the impact of repeated intermittent short sleep, with short sleep maintained 5 days per week followed by 2 days of prolonged sleep, compared to daily adequate sleep, on energy balance and cardiometabolic risk. A secondary goal of this research is to determine if maintaining a constant midpoint of sleep while undergoing intermittent short sleep, leads to better outcomes than intermittent short sleep with a 2-hour delay in sleep midpoint. The aims of this research will be tested in the context of a 3-group, parallel-arm, outpatient intervention of 4 weeks in duration, in young-to-middle-aged adults (aged 18-49 years).

DETAILED DESCRIPTION:
A large portion of the U.S. adult population reports insufficient sleep on a nightly basis. It has been shown that sustained insufficient sleep leads to adverse cardiometabolic risk profile and positive energy balance. However, sleep patterns in real life are not consistent over weeks. Individuals not obtaining sufficient sleep during the week may compensate by sleeping longer on weekends. The differences in sleep duration between week and weekend nights is approximately 1 hour, mostly due to delaying wake times rather than advancing bedtimes. A drawback of such behaviors is resultant change in sleep midpoint, which has been associated with adverse cardiometabolic health and obesity. However, very few studies have attempted to determine whether recovery sleep on weekends results in reversal of adverse health effects of insufficient sleep during the week. Available studies suggest that recovery sleep does not revert health markers to pre-sleep restriction (SR) levels. But these studies are short, usually involving only one cycle of SR followed by recovery sleep, and fail to use appropriate and robust statistical methods. Therefore, the goal of the current investigation is to evaluate the impact of repeated intermittent short sleep, with short sleep maintained 5 days/week followed by 2 days of recovery sleep, relative to daily adequate sleep, on energy balance and cardiometabolic risk markers. A secondary goal of this research is to determine if maintaining a constant sleep timing while undergoing intermittent short sleep, leads to better outcomes than intermittent short sleep in conjunction with shifts in sleep times.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 49 years
* BMI 20-29.9 kg/m2
* Habitually sleeping 7-9 hours/night without sleep aids or naps

Exclusion Criteria:

* Sleep disorders
* Psychiatric disorders (including eating disorders) and seasonal affective disorder
* Pregnancy (current/prior year)
* Breastfeeding
* Smokers (Any cigarette smoking or ex-smokers <3years)
* Diabetes
* Elevated blood pressure, taking beta-blockers
* Individuals taking anti-coagulants or anti-platelets
* Recent weight change or participation in a weight loss program or have ever had bariatric surgery or other weight loss or gastrointestinal procedure.
* Travel across time zones; shift work (non-traditional hours)

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2023-09-22 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Fasting Plasma Glucose | Up to 4 weeks
  Insulin resistance will be assessed by measuring fasting plasma glucose levels.
Insulin Level | Up to 4 weeks
  Insulin resistance will be assessed by measuring insulin levels.
Morning Systolic and Diastolic Blood Pressure | Up to 4 weeks
  Ambulatory blood pressure will be measured.
Evening Systolic and Diastolic Blood Pressure | Up to 4 weeks
  Ambulatory blood pressure will be measured.
Fat mass | Up to 4 weeks
  Body composition will be measured using Dual-energy X-ray absorptiometry (DXA) to determine fat mass.

SECONDARY OUTCOMES:
Low-density Lipoprotein (LDL) Level | Up to 4 weeks
  Lipid panel will be assessed.
High-density Lipoprotein (HDL) Level | Up to 4 weeks
  Lipid panel will be assessed.
Total Cholesterol Level | Up to 4 weeks
  Lipid panel will be assessed.
Triglyceride Level | Up to 4 weeks
  Lipid panel will be assessed.
C-reactive protein (CRP) Level | Up to 4 weeks
  CRP will be measured as an inflammatory marker.
Interleukin 6 (IL-6) | Up to 4 weeks
  IL-6 will be measured as an inflammatory marker.
Tumor necrosis factor alpha (TNF-alpha) | Up to 4 weeks
  TNF-alpha will be measured as an inflammatory marker.
Total daily energy expenditure | Baseline and endpoint (4 weeks)
  Energy expenditure will be measured using doubly-labeled water over 14 days
Energy Intake | Baseline and endpoint (4 weeks)
  Energy intake will be measured to assess diet quality using daily food records for 7 days.
Total Ghrelin | 2 hours post meal at baseline and endpoint (4 weeks)
  Total ghrelin will be assessed using radioimmunoassay (RIA).
Serum Leptin | 2 hours post meal at baseline and endpoint (4 weeks)
  Serum leptin will be measured using a double-antibody RIA.
Adiponectin Level | Up to 4 weeks
  Adiponectin levels will be analyzed using RIA.
Glucagon-like peptide 1 (GLP-1) Level | 2 hours post meal at baseline and endpoint (4 weeks)
  GLP-1 will be measured by RIA after plasma extraction with 95% ethanol.
Change in Nuclear factor kappa B (NFkB) Level | Baseline and endpoint (4 weeks)
  NFkB will be measured to assess endothelial cell inflammation.

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Pierre St-Onge, PhD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Data from this study will be available for sharing with other investigators. Data sharing requests should be made in writing and sent directly to the investigator(s) who generated the data. The purposes for using shared data should be stated in the request, and the data can only be used for research purposes. Data sharing agreements should be developed and accepted by both parties before data sharing takes place. Protecting the rights and privacy of human subjects and maintaining the study participants' confidentiality will be the first priority of our data sharing plan. HIPAA privacy rule for de-identification of a dataset will be followed before transferring data.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will become available after results of the main aims from the final dataset have been accepted for publication.
Access Criteria: Contact PI for information on data availability and data sharing.